CLINICAL TRIAL: NCT04387721
Title: Influence of Residual Astigmatism on Visual Acuity in Patients Undergoing Cataract Surgery With Trifocal Intraocular Lens Implantation
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Enrique Ordiñaga-Monreal, OD, MSc (Other)
Responsible Party: Sponsor-Investigator, Enrique Ordiñaga-Monreal, OD, MSc, Clinical Optometrist, Clinica Oftalmologica TACIR
Organization: Clinica Oftalmologica TACIR (Other)
Other Study IDs: EC042019; 2019/65-OFT-CMT (Other: CEIm Grupo Hospitalario Quirónsalud-Catalunya)
Record Dates: First submitted 2020-05-11; First posted 2020-05-14 (Actual); Last update posted 2020-05-14 (Actual); Status verified 2020-05

CONDITIONS: Cataract After; Astigmatism; IOL; Visual Acuity
Keywords: CSF; Contrast Sensitivity; Trifocal IOL
MeSH Terms: conditions — Capsule Opacification; Astigmatism

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Trifocal IOL(Finevision IOL, PhysIOL): We will divide the sample into two groups of patients depending on the IOL implanted First group: FineVision
  Interventions: Other: Kind of trifocal IOL
- Trifocal toric IOL (Finevision Toric IOL, PhysIOL): We will divide the sample into two groups of patients depending on the IOL implanted: Second group: FineVisionToric
  Interventions: Other: Kind of trifocal IOL

INTERVENTIONS:
Other: Kind of trifocal IOL — Patients will be divided between groups based on pre-surgery corneal astigmatism. Group FineVision is made up of patients with corneal astigmatism less than 1 D. Groups FineVision Toric is made up pf patients with corneal astigmatism more than 1.25 D
  Other Names: FineVision IOL; FineVision Toric IOL

SUMMARY:
MAIN OBJECTIVE: To assess the influence of residual astigmatism on visual acuity in the different lens foci in patients operated on for cataracts with a trifocal intraocular lens implant.

SECONDARY OBJECTIVE: To study the influence of residual astigmatism on the visual quality of the patient in the far focus and to determine if there are differences of affectation in the two study groups.

DETAILED DESCRIPTION:
It will be studied how small residual astigmatisms after cataract surgery degrade the visual acuity of patients in the three focal planes of trifocal IOLs. Not only VA will be studied, but also visual quality through contrast sensitivity curves.

ELIGIBILITY:
Inclusion Criteria:

* Bilateral surgery performed by the same surgeon
* IOLs implanted IOLs FineVision (MicroF) and FineVision Toric (PodFT)
* Patients with pre-surgery corneal astigmatism less than 2.5 D
* Patients whose pupillary diameter in physiological position (conditions of lower photopic pupil) not over 4 mm.

Exclusion Criteria:

* Post-surgical refractive residual astigmatisms ≧ 1.55D
* Previous corneal or intraocular surgeries
* Active diseases
* Eye complications during the 3-month follow-up

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The field in which it will carry out the study is a private medical centre. TACIR Ophthalmology clinic is located in the TEKNON Medical Center in the city of Barcelona. The study population will be the patients of the TACIR ophthalmology clinic who will be operated on cataracts and agree to take part in the study.
Sampling Method: Probability Sample
Enrollment: 48 (Estimated)
Dates: Start 2019-07-29 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2021-07 (Estimated)

PRIMARY OUTCOMES:
Visual Acuity | 3 months following cataract surgery
  Visual acuity will be measured at distance, intermediate distance (67 cm) and near (40 cm). Visual acuities will be obtained with logarithmic notation
Contrast Sensitivity Function (CSF) | 3 months following cataract surgery
  Contrast sensitivity will be measured at far, intermediate distance (67 cm) and near (40 cm).

SECONDARY OUTCOMES:
Differences between groups | 3 months following cataract surgery
  Results will be compared between groups.

CONTACTS AND LOCATIONS:
Overall Officials: Enrique Ordiñaga-Monreal, OD, Principal Investigator — Clinica Oftalmologica TACIR
Locations (1):
- Clinica Oftalmológica TACIR, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Statistical Analysis Plan (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04387721/SAP_000.pdf
  • Informed Consent Form (2019-07-29): https://cdn.clinicaltrials.gov/large-docs/21/NCT04387721/ICF_001.pdf